CLINICAL TRIAL: NCT02559973
Title: A Single-Center, Randomized, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Depot Buprenorphine (RBP-6000) Using Poly (DL-lactide-co-glycolide) Polymer of Two Different Molecular Weights (Low and High Molecular Weights as Test Treatments) in Comparison to Intermediate Molecular Weight (Reference Treatment) in Treatment-Seeking Subjects With Opioid Use Disorder
Brief Title: Pharmacokinetics, Safety, and Tolerability of Depot Buprenorphine at Three Different Molecular Weights in Treatment-Seeking Subjects With Opioid Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-13-0006
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Opioid Use Disorder
Keywords: Buprenorphine; opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- RBP-6000 - Light MW (Experimental): Single subcutaneous injection of RBP-6000 (buprenorphine) 300 mg, formulated with a light molecular weight (MW) polymer.
  Interventions: Drug: RBP-6000; Drug: SUBOXONE Sublingual Film
- RBP-6000 - Heavy MW (Experimental): Single subcutaneous injection of RBP-6000 (buprenorphine) 300 mg, formulated with a heavy molecular weight (MW) polymer.
  Interventions: Drug: RBP-6000; Drug: SUBOXONE Sublingual Film
- RBP-6000 - Intermediate MW (Active Comparator): Single subcutaneous injection of RBP-6000 (buprenorphine) 300 mg, formulated with an intermediate molecular weight (MW) polymer (reference).
  Interventions: Drug: RBP-6000; Drug: SUBOXONE Sublingual Film

INTERVENTIONS:
Drug: RBP-6000 — RBP-6000 uses buprenorphine in the ATRIGEL Delivery System. The single-syringe is prefilled with RBP-6000 containing 300 mg buprenorphine.
  Other Names: buprenorphine
Drug: SUBOXONE Sublingual Film — Subjects will be dose-stabilized on SUBOXONE sublingual film prior to administration of RBP-6000. SUBOXONE sublingual film will be administered beginning after the subject is experiencing signs and symptoms of withdrawal on Day -8 and continue until Day -1.
  Other Names: buprenorphine HCl and naloxone HCl dihydrate

SUMMARY:
This is a single-center, randomized, open-label, single-dose, parallel-group study which will enroll and randomize approximately 48 subjects (to achieve 36 completers) with opioid use disorder (OUD) who are seeking treatment for OUD. The study includes both a Residential (Inpatient) and Non-Residential (Outpatient) Period.

ELIGIBILITY:
Inclusion Criteria:

* Currently meets DSM-5 criteria for moderate or severe opioid use disorder (OUD)
* Is seeking treatment for OUD
* Body mass index: ≥ 18.0 to ≤ 35.0 kg/m^2
* Females: Female individuals of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to informed consent) must have a negative serum pregnancy test prior to enrollment and must agree to use a medically acceptable means of contraception from Screening through at least 6 months after the last dose of Investigational Medicinal Product (IMP).
* Males: Male individuals with female partners of child-bearing potential must agree to use medically acceptable contraception after signing the informed consent form through at least 6 months after the last dose of IMP. Male individuals must also agree not to donate sperm during the study and for 6 months after receiving the last dose of IMP.
* Have a normal electrocardiogram (ECG) or ECG with no clinically significant findings in the opinion of the Investigator or medically qualified sub-investigator at Screening and through pre-dose on Day 1.
* Agree not to take any buprenorphine-containing products, other than those administered for the current study, throughout the duration of the study.
* Willing to adhere to study procedures and provide written informed consent prior to start of any study procedures.

Exclusion Criteria:

* Current diagnosis, other than OUD, requiring chronic opioid treatment.
* Pregnant or lactating females.
* Have an ECG demonstrating a corrected QT interval using Fridericia's calculation (QTcF) > 450 msec in males and QTcF > 470 msec in females upon admission to the residential facility or prior to administration of RBP-6000.
* Currently meet the criteria for diagnosis of moderate or severe substance use disorder, by DSM-5 criteria, for any substances other than opioids, and/or tobacco.
* Had a significant traumatic injury, major surgery, or open biopsy within the 4 weeks prior to signing the informed consent form.
* Used buprenorphine-containing products within the 14 days prior to signing the informed consent form.
* Have a history of suicidal ideation within the 30 days prior to signing the informed consent form or prior to study drug administration
* Have a history or presence of allergic or adverse response (including rash or anaphylaxis) to buprenorphine, naloxone, methadone, or the ATRIGEL Delivery System.
* Individuals who have a positive urine drug screen (UDS) prior to admission to the residential facility for barbiturates, benzodiazepines, buprenorphine, or methadone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Study Day 1 to Day 29 (AUC0-28days) of Buprenorphine | Day 1 to Day 29
  Relative bioavailability will be assessed using AUC0-28days.
Maximum Observed Plasma Concentration (Cmax) of Buprenorphine | Day 1 to Day 57
  Relative bioavailability will also be assessed using Cmax

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Study Day 1 to Day 29 (AUC0-28days) of Norbuprenorphine | Day 1 to Day 29
Maximum Observed Plasma Concentration (Cmax) of Norbuprenorphine | Day 1 to Day 57
Participants with Treatment-Emergent Adverse Events | Day 1 to Day 57

CONTACTS AND LOCATIONS:
Locations (1):
- Vince & Associates Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No